CLINICAL TRIAL: NCT05091580
Title: The Effectiveness and Cost-effectiveness of Implementing Evidence-based Depression Treatment Within the TB Care Platform in South Africa: A Hybrid Effectiveness-implementation Trial
Brief Title: Effectiveness and Cost-Effectiveness of Depression Treatment for Individuals With TB in South Africa
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Interruption in funding
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); Desmond Tutu HIV Foundation (Other); University of Cape Town (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Annika Sweetland, Assistant Professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8217; R01AI148461 (NIH)
Record Dates: First submitted 2021-09-28; First posted 2021-10-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Depression; Tuberculosis
Keywords: effectiveness; cost-effectiveness; implementation science; Hybrid Type I Trial; South Africa; Depression; Tuberculosis
MeSH Terms: conditions — Depression; Tuberculosis

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized hybrid type I effectiveness-implementation trial
Masking Description: Since this is a stepped wedge design, masking will not be possible. Clinics will be randomized in terms of the order in which they're trained to deliver the behavioral intervention over time, but it will be obvious whether or not a clinic is implementing the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Interpersonal Counseling for Depression (Experimental): New adult TB patients with depressive symptoms (PHQ-9 > 10) will be offered 4-8 sessions of Interpersonal Counseling delivered by a trained lay counsellor.
  Interventions: Behavioral: Interpersonal Counseling
- Control: Enhanced Treatment as Usual (Other): New adult TB patients will be screened for depression and those with significant symptoms (PHQ-9 > 15 and/or suicidal ideation) will be referred to the clinic nurse for evaluation and referral to specialized mental health care as needed. Routine screening for depression is not a standard practice for TB patients; therefore assessment and referral is considered "enhanced" treatment as usual. Individuals will be interviewed at baseline and treatment completion.
  Interventions: Behavioral: Enhanced treatment as usual

INTERVENTIONS:
Behavioral: Interpersonal Counseling — Interpersonal Counseling is a brief (4-8 sessions) psychological intervention that was developed to treat depression in primary care. In IPC, counselors provide psychoeducation about the connection of depressive symptoms to social triggers and support patients in leveraging social networks to address these stressors and reduce depressive symptoms. Since depressive symptoms are often a transient reaction to life stress (e.g. TB diagnosis), many individuals are able to achieve significant alleviation of symptoms in as few as four sessions. IPC focuses on reducing interpersonal conflict and improving social cohesion in families, which may have the advantage of strengthening the ability of families to support TB patients in completing treatment to achieve cure. All individuals will be offered 4-5 sessions (weekly), with up to 3 optional booster sessions (monthly) until TB treatment is completed.
  Arms: Intervention: Interpersonal Counseling for Depression
Behavioral: Enhanced treatment as usual — Depression screening and referral (as needed)
  Arms: Control: Enhanced Treatment as Usual

SUMMARY:
This hybrid type I effectiveness-implementation trial will increase understanding of the effectiveness and cost-effectiveness of integrating a brief evidence-based treatment for major depressive disorder (MDD) within the tuberculosis (TB) care platform to improve TB and MDD. Findings from this R01 are likely to inform policy and treatment guidelines for the integrated management of TB and MDD in low- and middle-income countries globally.

DETAILED DESCRIPTION:
TB and depression are the leading infectious cause of death and the leading cause of disability, respectively. Furthermore, they are commonly co-occurring and negatively synergistic. TB and depression comorbidity is associated with a 2.85 greater chance of death and 8.70 higher risk for loss to follow up (LTFU) from treatment, which has a cascade of negative individual-, community-, societal-, and health system-level implications. As a treatable condition, depression is a remediable driver of the TB epidemic. The WHO has called for a global policy framework for TB and mental health integration, recommending brief psychological interventions to address mental disorders in primary care settings. Interpersonal counseling (IPC) is a brief version of one such evidence-based intervention that has demonstrated efficacy and effectiveness in treating depression when delivered by non-mental health specialists, including in South Africa. The purpose of this study is to assess the effectiveness and cost-effectiveness of integrating IPC (for depression) into the TB care platform to improve TB and depression outcomes, as well as mitigate TB-related catastrophic costs. As the country with the highest TB burden in the world, nearly 60% of whom are co-infected with HIV, South Africa is the ideal setting for this study. This 3-year hybrid type I effectiveness-implementation trial will be implemented in eight clinics (n~1410 individuals with TB/depression) in the Eastern and Western Capes of South Africa to integrate IPC to treat depression comorbidity within the TB care platform with the following aims: Aim 1) To evaluate the effectiveness and implementation outcomes of integrating IPC treatment for depression into the existing TB care platform to improve TB and depression outcomes; Aim 2) To determine the influence of theoretically based intervention mediators and moderators on TB treatment outcomes; Aim 3) To assess the cost-effectiveness of integrating depression treatment into the TB care platform from the patient and health system perspectives. This research will provide critical clinical, programmatic, and economic data to inform the WHO global policy framework for TB and mental health integration, and cost-effective clinical practice to improve TB outcomes, especially in low-resource settings.

Recruitment was temporarily paused on September 1, 2024 due to an interruption in funding.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* initiating treatment for TB
* ability to provide informed consent

Exclusion Criteria:

* unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
TB treatment success rate | 6 months
  Patient level TB treatment success (yes/no) will be extracted from clinic records and defined based on the South African National TB Control Guidelines as all smear-positive patients that were cured (negative smear in last month of treatment) and those that completed treatment but did not meet the criteria for cure or failure.

SECONDARY OUTCOMES:
Depression remission rate | 2 months, 6 months
  Patient level depression remission (yes/no) will be assessed using the Patient Health Questionnaire (PHQ-9) and defined as a score less than 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Desmond Tutu HIV Foundation, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Sharing of scientific findings with the research and clinical communities will be executed through the centralized NIH data repository, publications in peer reviewed journals, and presentations at scientific meetings. If requested, we will share our statistical code (SAS, Stata, R) for use with other investigators. We will also post the methods and analysis plan of this proposal on the Open Science Framework hosted by the Center for Open Science. Data to be shared will include all of the individual participant data collected during the trial, after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.